CLINICAL TRIAL: NCT01038141
Title: Recto Anal Repair or Milligan Morgans Operation of Grade 3 and 4 Symptomatic Haemorrhoidal Disease. A Prospective Randomized Controlled Study
Brief Title: Recto Anal Repair or Milligan Morgans Operation of Grade 3 and 4 Symptomatic Haemorrhoidal Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to lack of time.
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Geir Arne Larsen, M.D., Ph.D., Akershus University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 583-07315a 1.2007.2484(REK)
Record Dates: First submitted 2009-12-22; First posted 2009-12-23 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-06

CONDITIONS: Symptomatic Haemorrhoidal Disease
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Milligan Morgan (Active Comparator)
  Interventions: Procedure: Surgery for advanced haemorrhoidal disease
- Recto Anal Repair (Active Comparator)
  Interventions: Procedure: Surgery for advanced haemorrhoidal disease

INTERVENTIONS:
Procedure: Surgery for advanced haemorrhoidal disease — Milligan Morgan vs Recto Anal Repair
  Other Names: Transanal doppler-guided hemorrhoidal artery ligation.; Transanal hemorrhoidal dearterialization (THD).

SUMMARY:
The purpose of this study is to compare a new mini invasive surgical procedure (Recto Anal Repair) to the traditional Milligan-Morgan procedure in patients suffering from severe piles.

DETAILED DESCRIPTION:
An estimated 4% of the adult population suffers from haemorrhoidal disease. In 1937 E. T. Milligan and C. N. Morgan described a method for operating piles that still is regarded "the gold standard" in the treatment of severe haemorrhoidal disease. This procedure is followed by a prolonged and painful recovery. To overcome the long recovery often combined with long sick leaves, less invasive methods for treating piles have been introduced during the last decade. However, few studies have compared patient benefits and the long term outcome of these techniques, and the choice of treatment is often based on the skills and experience of the individual surgeon. A new and promising mini invasive approach utilizes doppler-guided ligation of the haemorrhoidal arteries. All haemorrhoidal arteries are identified and then ligated approximately 2 cm above the anal canal. Thereafter the rectal mucosa with the piles is repositioned and fixed in the rectum with running sutures. This procedure is termed Recto Anal Repair (RAR) and leads to shrinking of the piles and restored anatomy of the anus and the rectum. The investigators want to execute a randomized, consecutive, prospective, controlled study with long term follow up to compare the RAR procedure to Milligans operation for the treatment of severe haemorrhoidal disease.

The primary goals are evaluation of pain and sick leave 7, 14 and 21 days after surgery and reported reduction of pile symptoms after 3, 6 and 12 months. In addition the investigators want to compare the overall satisfaction with the two procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic grade 3 and 4 haemorrhoidal disease
* Age 18-80
* Patients who are fitted for local and general anaesthesia
* Patients who are able to understand the information given and are willing to give a written consent

Exclusion Criteria:

* Previous operated for piles
* Previous operated in the anal canal
* Faecal incontinence
* Inflammatory bowel disease with affection of the anal canal
* Chronic diarrhea
* Fissura ani
* Fistula in ano
* Chronic anal pain
* Neurological illness with affection of anal sensation
* Patients not able to follow the study protocol
* Patients taking immunosuppressant medication
* Pregnancy
* Disability
* Anal polyps
* Medication affecting the coagulation system
* Circular anal prolapse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-11; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain | up to 21 days

SECONDARY OUTCOMES:
Evaluation of sick leave | up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Geir A Larsen, M.D., Ph.D., Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lorenskog, Norway